CLINICAL TRIAL: NCT04046445
Title: An Open-Label, Multicenter, Non-Randomized, Dose-Confirmation and Cohort-Expansion Phase 1b Study to Evaluate the Safety, Tolerability, and Anti-Tumor Activity of ATP128, VSV-GP128 and BI 754091, in Patients With Stage IV Colorectal Cancer
Brief Title: Phase 1b Study to Evaluate ATP128, VSV-GP128 and BI 754091, in Patients With Stage IV Colorectal Cancer
Acronym: KISIMA-01
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Amal Therapeutics (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KISIMA-01; 2019-000728-16 (EudraCT Number); 2021DR1011 (Other: Swissmedic)
Record Dates: First submitted 2019-07-30; First posted 2019-08-06 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Colorectal Cancer; MSS; Stage IV Colon Cancer; Stage IV Rectal Cancer; Metastatic Colorectal Cancer; Liver Metastasis Colon Cancer
Keywords: CRC; Colorectal Cancer; MSS; Metastatic Colorectal Cancer; Liver Metastasis Colon Cancer; Stage IV Colon Cancer; Stage IV Rectal Cancer; KISIMA-01; ATP128; BI 754091 (Ezabenlimab); MMRp; VSV-GP128; Therapeutic viral vaccine; Heterologous prime-boost; Maintenance setting
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: 8 cohorts
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cohort 1a (Experimental): 6 patients with stage IV CRC who failed SoC therapies
  Interventions: Drug: ATP128
- Cohort 1b (Experimental): 6 patients with stage IV MSS/MMRp CRC in SD or PR after first line of SoC
  Interventions: Drug: ATP128; Drug: BI 754091
- Cohort 2a (Experimental): 5 patients with stage IV MSS/MMRp CRC in SD or PR after first line of SoC
  Interventions: Drug: ATP128; Drug: BI 754091
- Cohort 2b (Experimental): 15 patients with stage IV MSS/MMRp CRC with liver-limited disease
  Interventions: Drug: ATP128; Drug: BI 754091
- Cohort 2c (Experimental): 19 patients with stage IV MSS/MMRp CRC in SD or PR after first line of SoC
  Interventions: Drug: ATP128; Drug: BI 754091
- Cohort 3 (Experimental): 6 patients with stage IV MSS/MMRp CRC in SD or PR after first line of SoC
  Interventions: Drug: ATP128; Drug: BI 754091; Drug: VSV-GP128
- Cohort 4a (Experimental): 24 patients with stage IV MSS/MMRp CRC in SD or PR after first line of SoC
  Interventions: Drug: ATP128; Drug: BI 754091; Drug: VSV-GP128
- Cohort 4b (Experimental): 15 patients with stage IV MSS/MMRp CRC with liver-limited disease
  Interventions: Drug: ATP128; Drug: BI 754091; Drug: VSV-GP128

INTERVENTIONS:
Drug: ATP128 — 5-6 SC injections
Drug: BI 754091 — ≥ 7 IV infusions
  Other Names: Ezabenlimab
  Arms: Cohort 1b; Cohort 2a; Cohort 2b; Cohort 2c; Cohort 3; Cohort 4a; Cohort 4b
Drug: VSV-GP128 — 1 single IV injection
  Arms: Cohort 3; Cohort 4a; Cohort 4b

SUMMARY:
This is a multi-center, non-randomised Phase 1b study to evaluate the safety and tolerability of ATP128 alone or in combination with BI 754091 and of heterologous prime-boost ATP128 + VSV-GP128 in combination with BI 754091.

ATP128 is a self-adjuvanted chimeric recombinant protein vaccine being developed in combination with programmed cell death 1 (PD-1) blockade for the treatment of microsatellite stable (MSS) patients not responding to PD-1 blockade. The PD-1 inhibitor being tested with ATP128 is the BI 754091 (Ezabenlimab) compound which belongs to the human immunoglobulin G4 (IgG4) subclass of antibodies.

VSV-GP is a recombinant chimeric vesicular stomatitis virus (VSV, Indiana strain Rhabdoviridae) which carries the envelope glycoprotein (GP) of the visceral non neurotropic WE-HPI strain of the Lymphocytic choriomeningitis virus (LCMV, Arenaviridae) instead of the native VSV glycoprotein (G) and is developed as integral part of the prime-boost regimen together with ATP128.

The Sponsor plans to enrol 96 patients with histologically or cytologically confirmed stage IV colorectal cancer coming form three different patient populations:

* Cohort 1a: 6 patients with stage IV colorectal cancer (CRC) having failed standard of care (SoC) therapies
* Cohorts 1b, 2a, 2c: 30 patients with stage IV microsatellite stable/mismatch repair-proficient (MSS/MMRp) CRC being in stable disease (SD) or partial response (PR) after first line of SoC (4-6 months duration at minimum)
* Cohorts 2b, 4b: 30 patients with stage IV MSS/MMRp liver-limited disease

Patients eligible for this study will be enrolled in one of the 8 cohorts depending on their disease:

* Patients in Cohort 1a will receive ATP128 as single agent
* Patients in Cohorts 1b, 2a, 2b, 2c will receive ATP128 in combination with BI 754091
* Patients in Cohorts 3, 4a, 4b will receive ATP128 and VSV-GP128 in combination with BI 754091

ELIGIBILITY:
Inclusion Criteria:

Cohort 1a

1. Ability to comprehend and willingness to provide written informed consent (ICF) for the study.
2. Age ≥ 18 years.
3. Patient with histologically or cytologically confirmed stage IV CRC who has failed standard therapies.
4. Must have received Standard of Care systemic treatment consisting of fluoropyrimidin- oxaliplatin and/or irinotecan based therapy for stage IV CRC disease.
5. Presence of at least 1 measurable lesion by computed tomography or magnetic resonance imaging per RECIST v1.1 as determined by the local site investigator/radiologist assessment.
6. Presence of at least one liver lesion amenable to repeated biopsy, ideally not the one being used for measuring.
7. Willingness to undergo two fresh liver biopsies (pre-treatment and on-treatment).
8. Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.
9. Life expectancy of at least 3 months.
10. Resolution of all toxicities and any toxic effect(s) of the most recent prior therapy to Grade 1 or less (except alopecia). Patients with ≤ Grade 2 neuropathy and Grade ≤ 2 fatigue are an exception and may enroll.
11. Adequate renal, hepatic, and hematologic functions as defined by laboratory parameters ≤ 7 days before study treatment initiation.
12. Absolute neutrophil count (ANC) ≥ 1.5 × 109/L.
13. Absolute lymphocyte count ≥ 0.5 × 109/L.
14. Platelets ≥ 100 × 109/L.
15. Hemoglobin level ≥ 9 g/dL.
16. Measured or calculated creatinine clearance (glomerular filtration rate can also be used in place of creatinine clearance) ≥ 50 mL/min according to the formula of Cockcroft-Gault.
17. Total bilirubin ≤ 1.5 × upper limit of normal (ULN); if total bilirubin is > 1.5 x ULN then direct bilirubin must be ≤ 1.5 × ULN. Patients with known Gilbert's Syndrome may enroll if total bilirubin ≤ 3 × ULN.
18. Alanine aminotransferase/aspartate aminotransferase (ALT/AST) ≤ 2.5 × ULN or ≤ 5 x ULN in patients with hepatic involvement.
19. A female patient is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

    Not a woman of childbearing potential (WOCBP) OR A WOCBP who agrees to use highly effective contraceptive methods during the treatment period and for at least 180 days after the last dose of study treatment and refrain from egg donation during this period.
20. A male patient must agree to use a contraceptive during the treatment period and for at least 180 days after the last dose of study treatment and refrain from donating sperm during this period.

Cohorts 1b, 2a, 2c, 3 and 4a:

1. Ability to comprehend and willingness to provide written informed consent (ICF) for the study.
2. Age ≥ 18 years.
3. Histologically or cytologically confirmed CRC and MSS/MMR proficient status confirmed by polymerase chain reaction (PCR)/ immunohistochemistry or next generation sequencing (NGS) assay at local institution.
4. Must have received a first line of SoC systemic therapy (physician choice) for stage IV disease and completed the therapy. They must have an ongoing partial response (PR) or a stable disease (SD) at the completion of this therapy, completion of therapy as defined by the investigator, however, with a minimum number of 4 months.

   Note: Patient may have also received prior adjuvant therapy for stage II or III colorectal cancer, however the adjuvant treatment for stage II and III will not be considered as a prior line of therapy in case of relapse more than 6 months after the end of treatment.
5. Presence of at least 1 measurable lesion by computed tomography or magnetic resonance imaging per RECIST v1.1 as determined by the local site investigator/radiologist assessment.
6. Presence of at least one metastatic lesion amenable to paired biopsies (same lesion to be biopsied twice, at baseline and on D36), ideally not the one being used for measuring. However, liver lesions must be prioritized. Non-liver metastatic lesion biopsies may be collected only if the patient has no liver lesion or if the liver lesion is not amenable to paired biopsies (e.g. due to its size or location) or if the liver biopsy represents a risk or an undue inconvenience for the patient health/condition per Investigator judgment. In such cases, where a patient has no lesion amenable to biopsy at all, the paired biopsies may be waived by the Sponsor on a case-by-case basis.
7. Willingness to undergo two biopsies (liver lesion must be prioritized). If the Investigator judges the biopsies to be a risk or an undue inconvenience for the patient health/condition, they may be waived by the Sponsor on a case-by-case basis.
8. ECOG performance status 0 to 2.
9. Life expectancy of at least 6 months.
10. Has resolution of all toxicities and any toxic effect(s) of the most recent prior therapy to Grade 1 or less (except alopecia). Patients with ≤ Grade 2 neuropathy and Grade ≤ 2 fatigue are an exception and may enroll.
11. Adequate renal, hepatic, thyroid and hematologic functions as defined by laboratory parameters ≤ 7 days before study treatment initiation.
12. Absolute neutrophil count ≥ 1.5 × 109/L.
13. Absolute lymphocyte count ≥ 0.5 × 109/L.
14. Platelets ≥ 100 × 109/L.
15. Hemoglobin level ≥ 9 g/dL.
16. Measured or calculated creatinine clearance (glomerular filtration rate can also be used in place of creatinine clearance) ≥ 50 mL/min according to the formula of Cockcroft-Gault (see Appendix 6).
17. Total bilirubin ≤ 1.5 × ULN; if total bilirubin is > 1.5 x ULN then direct bilirubin must be ≤ 1.5 × ULN. Patients with known Gilbert's Syndrome may enroll if total bilirubin ≤ 3 × ULN.
18. ALT/AST ≤ 2.5 × ULN or ≤ 5 × ULN in patients with hepatic involvement.
19. A female patient is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

    Not a woman of childbearing potential (WOCBP) OR A WOCBP who agrees to use highly effective contraceptive methods during the treatment period and for at least 180 days after the last dose of study treatment and refrain from egg donation during this period.
20. A male patient must agree to use a contraceptive during the treatment period and for at least 180 days after the last dose of study treatment and refrain from donating sperm during this period.

Specific to Cohorts 3, 4a, 4b:

1. Patient agrees to follow the instructions and precautions (see Section 4.4.1) related to potential VSV-GP128 shedding.

Cohorts 2b and 4b:

1. Ability to comprehend and willingness to provide written informed consent (ICF) for the study.
2. Age ≥ 18 years.
3. Histologically or cytologically confirmed CRC and MSS/MMR proficient status confirmed by PCR/immunohistochemistry or NGS assay at local institution.
4. Radiological evidence (CT/MRI) of liver-limited stage IV CRC.
5. Must have received first line neoadjuvant SoC systemic therapy (physician choice) for stage IV disease. May have received up to 16 weeks of this systemic SoC therapy.

   Note: Patient may have also received prior adjuvant therapy for stage II or III colorectal cancer, however the adjuvant treatment for stage II and III will not be considered as a prior line of therapy in case of relapse more than 6 months after the end of treatment.
6. Absence of disease progression following neoadjuvant chemotherapy.
7. Eligible for R0 complete liver metastasectomy (in case the primary tumor was already removed) or for R0 complete simultaneous combined resection (resection of both liver metastases and primary tumor in case the primary tumor is still in place) with curative intent.
8. ECOG performance status 0 to 2.
9. Life expectancy of at least 12 months.
10. Adequate renal, hepatic, thyroid and hematologic functions as defined by laboratory parameters ≤ 7 days before study treatment initiation.
11. Absolute neutrophil count ≥ 1.5 × 109 /L.
12. Absolute lymphocyte count ≥ 0.5 × 109 /L.
13. Platelets ≥ 100 × 109/L.
14. Hemoglobin level ≥ 9 g/dL.
15. Measured or calculated creatinine clearance (glomerular filtration rate can also be used in place of creatinine clearance) ≥ 50 mL/min according to the formula of Cockcroft-Gault (see Appendix 6).
16. Total bilirubin ≤ 1.5 × ULN; if total bilirubin is > 1.5 x ULN then direct bilirubin must be ≤ 1.5 × ULN. Patients with known Gilbert's Syndrome may enroll if total bilirubin ≤ 3 × ULN.
17. ALT/AST ≤ 2.5 × ULN or ≤ 5 × ULN in patients with hepatic involvement.
18. A female patient is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

    Not a woman of childbearing potential (WOCBP) OR A WOCBP who agrees to use highly effective contraceptive methods during the treatment period and for at least 180 days after the last dose of study treatment and refrain from egg donation during this period.
19. A male patient must agree to use a contraceptive during the treatment period and for at least 180 days after the last dose of study treatment and refrain from donating sperm during this period.

Exclusion Criteria:

All Cohorts:

1. Unwilling or unable to follow protocol requirements or to give informed consent.
2. Gastro-intestinal bowel obstruction (partial or complete).
3. Participation in any other study with an investigational study drug or device requires Medical Monitor approval.
4. Prior monoclonal antibody within 4 weeks or 5 half-lives (whichever is shorter) before administration of study treatment with the exception of bevacizumab (Avastin®), cetuximab (Erbitux®) and panitumumab (Vectibix®) which may have been received within 15 days from initiation of study treatment. Supportive care (e.g. denosumab) may be used before and during study treatment.
5. Prior therapy with checkpoint inhibitors (anti-programmed death 1 (anti-PD-1), anti-programmed death-ligand 1 (anti-PD-L1), anti-cytotoxic T-lymphocyte-associated protein 4 (anti-CTLA-4)). Patients must not have received any investigational immunotherapy neither.
6. Prior chemotherapy or targeted small molecule therapy within 15 days from initiation of study treatment.
7. Prior radiotherapy within 2 weeks of enrolment or within 4 weeks of enrolment in the case of radiation to central nervous system (CNS), which requires ≥ 4-week washout. Patients must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis.
8. Major (according the Investigator's judgment) surgery within 12 weeks before enrolment.
9. Known additional malignancy that is progressing or requires active treatment, or history of other malignancy within 2 years of study entry with the exception of cured basal cell or squamous cell carcinoma of the skin, superficial bladder cancer, prostate intraepithelial neoplasm, carcinoma in situ of the cervix, ductal or lobular carcinoma in situ of the breast, or other non-invasive or indolent malignancy, or cancers from which the patient has been disease-free for > 1 year, after treatment with curative intent.
10. Immunosuppression including the continued use of systemic (at prednisone dose equivalent of > 10 mg) or topical steroids at or near the injection site (excluding inhaled and eye drop-containing corticosteroids) or the use of immunosuppressive agents for any concurrent condition. All other corticosteroids must be discontinued > 4 weeks prior to first study treatment administration.
11. Previous vaccination (either therapeutic and/or prophylactic) against mCRC.
12. Pregnant/nursing women or unwilling to comply with acceptable contraceptive methods during study course.
13. History of autoimmune disease including any active autoimmune disease except vitiligo or childhood asthma.
14. Dermatological disease requiring local immunosuppressive agent.
15. Chronic or concurrent active infectious disease requiring systemic antibodies, antifungal, or antiviral treatment.
16. Known medical history of human immunodeficiency virus (HIV) infection or known medical history of acquired immunodeficiency syndrome (AIDS). HIV testing is not required unless mandated by the local health authority.
17. Has known history of or is positive for hepatitis B (hepatitis B virus surface antigen [HBsAg] reactive) or hepatitis C (HCV RNA).

    Note: Testing must be performed to determine eligibility. - Hepatitis B virus DNA must be undetectable and HBsAg negative at screening visit.- Hepatitis C antibody testing is allowed for screening purposes in countries where HCV RNA is not part of standard of care. In these cases, HCV antibody positive patients will be excluded.- Patients who have had definitive treatment for HCV are permitted if HCV RNA is undetectable at screening visit.
18. Known active CNS metastasis and/or carcinomatous meningitis.
19. Known cerebral oedema.
20. Live vaccine received within 30 days before initiation of study treatment. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, yellow fever, rabies, Bacillus Calmette-Guérin, and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed. however, intranasal influenza vaccines (FluMist®) are live attenuated vaccines and are not allowed. COVID-19 vaccines that are not live vaccines are allowed before and during study treatment. However, a COVID-19 vaccination should not occur within ± 2 days of ATP128 study drug and ± 15 days of VSV-GP128 study drug.
21. History of allergy or hypersensitivity to any of the study drugs or study drug components.
22. Any condition in the judgment of the Investigator which makes the patient unsuitable for trial participation.

    Cohorts 1b, 2a, 2b, 2c, 3, 4a and 4b:
23. Has received more than 1 line of therapy for stage IV disease (neoadjuvant therapy in Cohort 2b counts as 1 line).
24. History of pneumonitis within the last 5 years.
25. Active interstitial lung disease (ILD)/pneumonitis or a history of ILD/pneumonitis requiring treatment with systemic steroids and/or whose pulse oximetry is less than 92% "on room air".
26. Any of the following cardiac criteria:

    * Mean resting corrected QT interval (QTc) > 470 msec.
    * Any clinically important abnormalities (as assessed by the Investigator) in rhythm, conduction, or morphology of resting ECGs, e.g., complete left bundle branch block, third degree heart block.
    * Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years old, or any concomitant medication known to prolong the QT interval (according to institutional guidelines).
    * Ejection fraction (EF) < 55% or the lower limit of normal of the institutional standard will be excluded. Only in cases where the Investigator (or the treating physician or both) suspects cardiac disease with negative effect on the EF will the EF be measured during screening using an appropriate method according to local standards to confirm eligibility (e.g. echocardiogram [ECHO], multi-gated acquisition scan [MUGA]. A historic measurement of EF no older than 6 months prior to first study treatment administration can be accepted provided that there is clinical evidence that the EF value has not worsened since this measurement in the opinion of the Investigator or the treating physician or both.

Specific to Cohorts 3, 4a, 4b:

1. Previous treatment with VSV-based agents.
2. Use of Tamoxifen within one month prior the initiation of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2019-07-22 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate safety and tolerability by measure of incidence of treatment-emergent adverse events (AEs) and serious adverse events (SAEs) graded using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 | 1 year
  Safety
valuate anti-tumor effect of study treatment by measure of Progression-free survival (PFS) | 6 months
  Based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1

SECONDARY OUTCOMES:
Evaluate anti-tumor effect of study treatment by measure of Overall Response (OR) | 1 year
  Based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Confirm recommended phase 2 dose (RP2D) of study treatment | 1 year
  Based on evaluation of AEs with the support of pharmacodynamics
Further evaluate anti-tumor effect of study treatment of Best Overall Response (BOR) | 1 year
  Based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Evaluate anti-tumor effect of study treatment by measure of Duration of Response (DoR) | 1 year
  Based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Evaluate anti-tumor effect of study treatment by measure of Progression Free Survival (PFS) | 1 year
  Based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
Evaluate anti-tumor effect of study treatment by measure of Relapse Free Survival (RFS) | 1 year
  Based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1

OTHER OUTCOMES:
Evaluate pharmacodynamic effects of study treatment | 4.5 months
  Immune-monitoring based on blood and tissue samples
Detect early signal of relapse in tumor-free patients with liquid biopsy | 6 months
  Monitoring of ctDNA detection in the plasma
Further evaluate anti-tumor effect of study treatment by measure of PFS | 1 year
  Based on immune Response Evaluation Criteria in Solid Tumors (iRECIST)
Assess shedding and viremia of VSV-GP128 | 1 month
  Based on PCR and TCID50 in biological fluids

CONTACTS AND LOCATIONS:
Overall Officials: Scott Kopetz, Principal Investigator — MD Anderson
Locations (12):
- United States (7):
  - Honor Health Institute, Scottsdale, Arizona
  - University of Southern California, Los Angeles, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - NYU Langone Health, New York, New York
  - Weill Cornell Medicine, New York, New York
  - Duke Cancer Institute, Durham, North Carolina
  - University of Texas, MD Anderson Cancer Center, Houston, Texas
- Belgium (2):
  - University Hospital Antwerpen, Edegem
  - University Hospital Leuven, Leuven
- University Medicine Mainz, Mainz, Germany
- Switzerland (2):
  - University Hospital Zurich, Zurich, Canton of Zurich
  - Geneva University Hospitals, Geneva

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Namdari H, Rezaei F, Heidarnejad F, Yaghoubzad-Maleki M, Karamigolbaghi M. Immunoinformatics Approach to Design a Chimeric CD70-Peptide Vaccine against Renal Cell Carcinoma. J Immunol Res. 2024 Jan 27;2024:2875635. doi: 10.1155/2024/2875635. eCollection 2024. PMID 38314087